CLINICAL TRIAL: NCT01358032
Title: Evaluating the Effectiveness of an In-home Self-management Intervention to Prevent Psychological Distress in Frail Older People Living in the Community
Brief Title: Evaluating an In-home Multicomponent Program to Manage Concerns About Falling in Frail Community Dwelling Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 07-3-064; ZonMw 120610001 (Other Grant/Funding Number: ZonMw 120610001)
Record Dates: First submitted 2011-05-17; First posted 2011-05-23 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Concerns About Falling; Aged
Keywords: Fear of falling; Cognitive behavioral therapy; Randomized controlled trial; Frailty; Accidental Falls
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive behavioral program (Experimental): an in-home cognitive behavioral program on managing concerns about falling and associated activity avoidance in frail community-dwelling older people facilitated by trained community nurses.
  Interventions: Behavioral: an in-home cognitive behavioral program
- Control group (No Intervention): no program, only care as usual

INTERVENTIONS:
Behavioral: an in-home cognitive behavioral program — The in-home cognitive behavioral program aims to learn older persons, living in the community, how to deal with concerns about falling and to increase physical, social and functional activity. The principles of cognitive restructuring are used for shifting maladaptive in adaptive attitudes with respect to falling as well as increasing self efficacy beliefs and feelings of control. The following themes are discussed during the program: concerns about falling, thoughts about falling, physical exercise, assert oneself, overcome personal barriers, recognizing fall-ty habits and managing concerns about falling. Duration of the program is 10 weeks with 7 individual sessions (3 home visits (60, 60 and 75 minutes, respectively) & 4 telephone contacts (35 minutes each). The program is facilitated by trained nurses qualified in the field of geriatrics and working for home care agencies.
  Arms: Cognitive behavioral program

SUMMARY:
The main objectives of this study are:

1. an effect evaluation of an in-home multicomponent cognitive behavioural program on concerns about falling and related avoidance of activity (primary outcomes), as well as disability, fall incidents (secondary outcomes) and several additional outcomes in frail community-dwelling older people,
2. a process evaluation of the feasibility of the program, with the following main outcomes: population reached, performance according to protocol, exposure and engagement, opinion on the program of participants and facilitators, perceived benefit or achievement, and experienced barriers and potential solutions, and
3. an economical evaluation on the impact of the program on healthcare utilization and related costs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years or over
* At least some concerns about falling
* At least some associated avoidance of activity
* Fair or poor perceived general health
* Living independently in the community
* Written informed consent

Exclusion Criteria:

* Cognitive impairment (a score of less than 4 on the Abbreviated Mental Test 4)
* Language or hearing problems that impede completing an interview by telephone
* Sight problems that impede completing the intervention
* Confinement to bed
* Waiting for nursing home admission
* Permanent use of a wheelchair

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 389 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
concerns about falling | baseline, 5 months and 12 months
  Falls Efficacy Scale International (FES-I)
avoidance of activities due concerns about falling | baseline, 5 months and 12 months
  Falls Efficacy Scale International Avoidance Behaviour (FES-IAB)

SECONDARY OUTCOMES:
disability | baseline, 5 months and 12 months
  Groningen Activity Restriction Scale (GARS)
number of falls | continuous registration during the course of the trial for a period of 1 year
  Fall calendar
catastrophic beliefs about falling | baseline, 5 months and 12 months
  Catastrophic beliefs about falling (CAFS)
perceived consequences of falling | baseline, 5 months and 12 months
  CoF - loss of functional independence subscale and damage to identity subscale
perceived control over falling | baseline, 5 months and 12 months
  Perceived control over falling (PCOF)
mastery | baseline, 5 months and 12 months
  Personal Mastery Scale
feelings of anxiety | baseline, 5 months and 12 months
  Subscale of the Hospital Anxiety and Depression Scale (HADS-A)
symptoms of depression | baseline, 5 months and 12 months
  Subscale of the Hospital Anxiety and Depression Scale (HADS-D)
social support interactions | baseline, 5 months and 12 months
  Social support interactions (SSL 12-I)
health-related quality of life | baseline, 5 months and 12 months
  SF-12 Health Survey

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Background] Dorresteijn TA, Rixt Zijlstra GA, Van Eijs YJ, Vlaeyen JW, Kempen GI. Older people's preferences regarding programme formats for managing concerns about falls. Age Ageing. 2012 Jul;41(4):474-81. doi: 10.1093/ageing/afs007. Epub 2012 Feb 23. PMID 22367355
- [Background] Dorresteijn TA, Zijlstra GA, Delbaere K, van Rossum E, Vlaeyen JW, Kempen GI. Evaluating an in-home multicomponent cognitive behavioural programme to manage concerns about falls and associated activity avoidance in frail community-dwelling older people: Design of a randomised control trial [NCT01358032]. BMC Health Serv Res. 2011 Sep 20;11:228. doi: 10.1186/1472-6963-11-228. PMID 21933436
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Kruisbrink M, Zijlstra GAR, Crutzen R, Dorresteijn TAC, Winkens B, Kempen GIJM. Participant Characteristics as Moderators of the Effects of Cognitive Behavioral Interventions on Concerns About Falling: Secondary Analyses of Two Randomized Controlled Trials. J Appl Gerontol. 2023 Aug;42(8):1877-1887. doi: 10.1177/07334648231165904. Epub 2023 Apr 6. PMID 37026185
- [Derived] Evers SMAA, Dorresteijn TAC, Wijnen BFM, van Haastregt JCM, Kempen GIJM, Zijlstra GAR. Economic evaluation of a home-based programme to reduce concerns about falls in frail, independently-living older people. Expert Rev Pharmacoecon Outcomes Res. 2020 Dec;20(6):641-651. doi: 10.1080/14737167.2019.1666714. Epub 2019 Sep 20. PMID 31502897
- [Derived] Dorresteijn TA, Zijlstra GA, Ambergen AW, Delbaere K, Vlaeyen JW, Kempen GI. Effectiveness of a home-based cognitive behavioral program to manage concerns about falls in community-dwelling, frail older people: results of a randomized controlled trial. BMC Geriatr. 2016 Jan 6;16:2. doi: 10.1186/s12877-015-0177-y. PMID 26739339
- [Derived] Dorresteijn TA, Rixt Zijlstra GA, Van Haastregt JC, Vlaeyen JW, Kempen GI. Feasibility of a nurse-led in-home cognitive behavioral program to manage concerns about falls in frail older people: a process evaluation. Res Nurs Health. 2013 Jun;36(3):257-70. doi: 10.1002/nur.21534. Epub 2013 Mar 26. PMID 23533013